CLINICAL TRIAL: NCT06188507
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of GSK3996401 Following Single and Multiple Ascending Doses of GSK4347859 in Healthy Participants
Brief Title: A First Time in Human Study to Evaluate the Safety and Tolerability of GSK3996401 Following Dosing With GSK4347859 in Healthy Participants
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: The trial was temporarily halted due to findings in new non-clinical studies necessitating further investigation.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 221220
Record Dates: First submitted 2023-12-19; First posted 2024-01-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Lupus; GSK4347859; GSK3996401; Safety; First time in human (FTiH); Pharmacokinetics; Healthy Participants
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Click here to enter text.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Part 1: Cohort 1-GSK4347859 or Placebo (Experimental): Participants in Part 1 Cohort 1 will receive a single dose level of GSK4347859 dose level 1 or placebo in treatment period 1, followed by GSK4347859 dose levels 2 and 3 or placebo in 3- period dose escalation design. Additionally, there will be an optional 4th treatment period with dose level 4. Followed by a wash out period of at least 7 days between each dose.
  Interventions: Drug: GSK4347859; Drug: Placebo
- Part 1: Cohort 2-GSK4347859 or Placebo (Experimental): Participants in Part 1 Cohort 2 will receive a single dose level of GSK4347859 dose level 5 or placebo in treatment period 1, followed by GSK4347859 dose levels 6 and 7 or placebo in 3- period dose escalation design. Additionally, there will be an optional 4th treatment period with dose level 8. Followed by a wash out period of at least 7 days between each dose.
  Interventions: Drug: GSK4347859; Drug: Placebo
- Part 2: Cohort 3-GSK4347859 or Placebo (Experimental): Participants in Part 2 Cohort 3 will receive 14 days of repeat doses of GSK4347859 dose level A or placebo.
  Interventions: Drug: GSK4347859; Drug: Placebo
- Part 2: Cohort 4-GSK4347859 or Placebo (Experimental): Participants in Part 2 Cohort 4 will receive 14 days of repeat doses of GSK4347859 dose level B or placebo.
  Interventions: Drug: GSK4347859; Drug: Placebo
- Part 2: Cohort 5-GSK4347859 or Placebo (Experimental): Participants in Part 2 Cohort 5 will receive 14 days of repeat doses of GSK4347859 dose level C or placebo.
  Interventions: Drug: GSK4347859; Drug: Placebo

INTERVENTIONS:
Drug: GSK4347859 — GSK4347859 will be administered
Drug: Placebo — Placebo will be administered

SUMMARY:
This is a first time in human (FTiH) study which means that this is the first time that GSK4347859 is given to humans. The study is designed to investigate the safety, tolerability, and concentration of GSK3996401 (the activated form of GSK4347859) in the blood following single ascending doses (Part 1) and multiple ascending doses (Part 2) of GSK4347859 in healthy participants. Part 1 consists of 2 planned cohorts with up to 4 treatment periods in each and is expected to have up to 8 dose levels. Part 2 will investigate 14 days of repeat dosing in 3 cohorts with 3 dose levels.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are overtly healthy.
* Participant has a confirmed positive vaccination status for severe acute respiratory syndrome-related Coronavirus (2 SARS-CoV-2) and, if study dosing is during Flu season, influenza vaccines administered at least 30 days prior to dosing in the study.
* Fitzpatrick skin type I, II or III (Part 2 only).
* Body weight greater than or equal to (≥) 50 kilogram (kg) and body mass index (BMI) within the range 18 -32 kilogram per meter square (kg/m^2) (inclusive).
* Male and female of non-childbearing potential.
* Capable of giving signed informed consent.

Exclusion Criteria:

* History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, psychiatric, or neurological disorders. - Abnormal blood pressure
* A clinically significant ECG abnormality at screening.
* Evidence of active or latent tuberculosis (TB).
* Symptomatic herpes zoster within 3 months prior to screening
* Alanine transaminase (ALT) >1 times upper limit of normal (ULN).
* Total bilirubin >1.5x ULN [isolated total bilirubin >1.5x ULN is acceptable if total bilirubin is fractionated and direct bilirubin <35- percentage (%)].
* History of malignancy.
* Participants with known Corona virus disease-2019 (COVID-19) positive contacts as per local/site Guidelines
* Prior moderate/severe COVID-19 infection requiring oxygen supplementation or admission to hospital.
* Live vaccine(s) within 1 month prior to screening or plan to receive such vaccines during the study.
* Past or intended use of over-the-counter or prescription medication including herbal medications within 7 days prior to dosing
* The participant has participated in a clinical trial and has received an investigational product within 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product and dosing.
* Current enrolment or past participation in this clinical study
* Presence of Hepatitis B surface antigen (HBsAg) at screening or within 3 months prior to first dose of study intervention
* Positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study intervention
* Positive hepatitis C Ribonucleic acid (RNA) test result at screening or within 3 months prior to first dose of study
* Positive pre-study drug/alcohol screen
* Regular use of known drugs of abuse, including tetrahydrocannabinol.
* Positive Human immunodeficiency virus (HIV) antibody test
* Positive smoke breathalyzer levels indicative of smoking history at screening and each in-house admission to the clinical research unit or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Estimated glomerular filtration rate (eGFR) of less than (<) 90 (millilitre/minute) mL/min/1.73 m2 and / or Urine Albumin Creatinine (UACR) of >30 milligram per gram (mg/g) at screening
* A positive confirmation of SARS-CoV-2 infection or signs and symptoms suggestive of SARS-CoV-2 at screening or pre-dose
* The participant has a phobia to needles
* An average weekly alcohol intake of > 14 units.

For Part 2:

* History of benign skin conditions including but not limited to photosensitivity, atopic dermatitis, chronic eczema, psoriasis, urticaria, vitiligo, post-inflammatory hyperpigmentation, or keloid or hypertrophic scaring that in the opinion of the Investigator would impact study participation.
* History or presence of excessive bleeding or coagulation disorders.
* History of adverse reaction to local anesthetic.
* The presence of widespread acne, freckles, naevi, tattoos, birthmarks, piercings, scarring or other skin variations within the proposed Ultraviolet B (UVB) exposure challenge area
* Direct UV exposure to the areas of the body to be studied within 2 weeks.
* Unable to refrain from exposure to extended and direct sunlight or use of artificial tanning devices, self-tanning products, sun blocking products or other topical products (including moisturizers and makeup) on the areas of the body to be studied.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Estimated)
Dates: Start 2024-01-12 (Actual); Primary Completion 2026-07-14 (Estimated); Study Completion 2026-07-14 (Estimated)

PRIMARY OUTCOMES:
Part 1 - Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to Day 15
Part 2 - Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to Day 30
Part 1 - Number of Participants with Clinically Significant Changes in Haematology | Up to Day 15
Part 2 - Number of Participants with Clinically Significant Changes in Haematology | Up to Day 30
Part 1 - Number of Participants with Clinically Significant Changes in Clinical Chemistry | Up to Day 15
Part 2 - Number of Participants with Clinically Significant Changes in Clinical Chemistry | Up to Day 30
Part 1 - Number of Participants with Clinically Significant Changes in Laboratory Values for Urinalysis | Up to Day 15
Part 2 - Number of Participants with Clinically Significant Changes in Urinalysis | Up to Day 30
Part 1 - Number of Participants with Clinically Significant Changes in Vital Signs | Up to Day 15
Part 2 - Number of Participants with Clinically Significant Changes in Vital Signs | Up to Day 30
Part 1 - Number of Participants with Clinically Significant Changes in 12 Lead Electrocardiogram Readings | Up to Day 15
Part 2 - Number of Participants with Clinically Significant Changes in 12 Lead Electrocardiogram Readings | Up to Day 30
Part 1 - Number of Participants with Clinically Significant Changes in 24 Hour Telemetry | Up to Day 2
Part 2 - Number of Participants with Clinically Significant Changes in 24 Hour Telemetry | Up to Day 15

SECONDARY OUTCOMES:
Part 1 - Maximum observed plasma concentration (Cmax) of GSK3996401 following administration of GSK4347859 | Up to Day 3
Part 1 - Time to maximum observed plasma concentration (Tmax) of GSK3996401 following administration of GSK4347859 | Up to Day 3
Part 1 - Apparent terminal half-life (t½) of GSK3996401 following administration of GSK4347859 | Up to Day 3
Part 1 - Area under the concentration-time curve from zero to last quantifiable concentration [AUC(0-t)] of GSK3996401 following administration of GSK4347859 | Up to Day 3
Part 1 - Area under the concentration-time curve from time zero to infinity [AUC(0-∞)] of GSK3996401 following administration of GSK4347859 | Up to Day 3
Part 1 - Area under the concentration-time curve over each dosing interval [AUC(0-tau)] of GSK3996401 following administration of GSK4347859 | Up to Day 3
Part 1 - Area under the concentration-time curve from time zero to 24 hours after dosing [AUC(0-24)] of GSK3996401 following administration of GSK4347859 | Up to Day 3
Part 1 - Observed trough concentrations (Ctrough) of GSK3996401 following administration of GSK4347859 | Up to Day 3
Part 2 - Cmax of GSK3996401 following administration of single and repeat doses of GSK4347859 | Up to Day 15
Part 2 - Tmax of GSK3996401 following administration of single and repeat doses of GSK4347859 | Up to Day 15
Part 2 - Area under the concentration-time curve from time zero to 24 hours after dosing [AUC(0-24)] of GSK3996401 following administration single and repeat doses of GSK4347859 | Up to Day 15
Part 2 - Observed trough concentrations (Ctrough) of GSK3996401 following administration of GSK4347859 | Up to Day 15
Part 2 - Area under the concentration-time curve over each dosing interval [AUC(0-tau)] of GSK3996401 following administration of GSK4347859 | Up to Day 15

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United Kingdom (2):
  - GSK Investigational Site, Cambridge
  - GSK Investigational Site, Nottingham

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/